CLINICAL TRIAL: NCT06697275
Title: Evaluation of the Efficacy of a Virtual Reality When Placing a Needle on an Implantable Venous Access Device in Children With Leukemia: Randomized Multicenter Trial
Brief Title: Evaluation of the Efficacy of a Virtual Reality When Placing a Needle on an Implantable Venous Access Device in Children With Leukemia
Acronym: LEAVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PHRIP-2022-USCLADE; 2023-A02154-41 (Other: ANSM)
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Virtual Reality; Children and Adolescents; Acute Leukemia; Anxiety and Fear
Keywords: acute leukemia; virtual reality mask; children and adolescents from 6 to 16
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, open-label, three arms parallel, multicenter therapeutic trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard method (Active Comparator): In this standard method, before the treatment, the procedure of inserting the needle into the implantable port is explained to the child. The patient is comfortably installed and the treatment start using the standard method which consist on distracting the patient by singing, story telling, talking etc..
  Use of local anesthesic cream and +/- anxiolytic gas
  Interventions: Other: Standard method
- Interactive virtual reality (Active Comparator): Before the treatment, the caregiver explains the procedure of inserting the needle into the implantable port. A general explanation is given on the VR device (how the headphones and headsets are placed), presentation of the virtual worlds to choose from, description of the course of the session (virtual travel is guided by a voice). For the interactive virtual reality, the mode of operation will be explained as the actions are validated using the eyes.
  The patient is then installed comfortably. The caregiver helps the child to put on the headphones and headset correctly. Before starting the care procedure, the caregiver will wait about 5 minutes after the start of the viewing to make sure the child is completely immersed in the virtual reality. The software is turned off about 3 minutes after the end of the care procedure.
  Use of local anesthesic cream.
  Interventions: Device: Interactive virtual reality
- Hypnotic virtual reality (Active Comparator): Before the treatment, the caregiver explains the procedure of inserting the needle into the implantable port to the child. A general explanation is given on the VR device (how the headphones and headsets are placed), presentation of the virtual worlds to choose from, description of the course of the session (virtual travel is guided by a voice). The patient is then installed comfortably. The caregiver helps the child to put on the headphones and headset correctly. Before starting the care procedure, the caregiver will wait about 5 minutes after the start of the viewing to make sure the child is completely immersed in the virtual reality. The software is turned off about 3 minutes after the end of the care procedure.
  Use of local anesthesic cream.
  Interventions: Device: Hypnotic Virtual reality

INTERVENTIONS:
Device: Hypnotic Virtual reality — Hypnotic Virtual reality mask Deepsen® with age-appropriate software Birdy®
  Arms: Hypnotic virtual reality
Device: Interactive virtual reality — Interactive virtual reality mask Deepsen® with age-appropriate software Birdy®
  Arms: Interactive virtual reality
Other: Standard method — Use of local anesthesic cream + Nurse and/or parents distraction +/- anxioloytic gas
  Arms: Standard method

SUMMARY:
Main objective:

Evaluate the effectiveness of the repeated use of interactive or hypnotic virtual reality compared to standard treatment, on pain, during each needle placement on PAC for 3 months on children or adolescents (6 to 16 years old) with acute leukemia

Hypothesis:

Repeated use over 3 months of hypnotic or interactive virtual reality provides more benefits in terms of :

* pain management
* anxiety of the child and his parents
* satisfaction of the child's care, of his parents and of the caregivers compared to the standard method when inserting a needle into an implantable port in the pediatric oncology department or day hospital.

DETAILED DESCRIPTION:
Children and adolescents with acute leukemia frequently have anxiety-provoking and painful care in the management of their disease. As soon as the diagnosis is announced, the installation of a central line is recommended to allow the administration of chemotherapy treatments, parenteral nutrition, and blood tests. The implantable port (IP) is more often used than the central catheter. It allows the injection of drugs directly into the implantable port, through the skin using a specific needle whose caliber can be variable. This treatment, which can be repeated weekly, causes pain and anxiety for children. The use of skin anesthetic patches (EMLA®) is recommended to limit pain during needle installation. According to the literature, this system limits the pain associated with needle injections but does not reduce children's anxiety about this upcoming treatment. The repetition of the gesture, often for several months, is a source of discomfort and pain that only increases over time. A memorization of pain increases the apprehension of care by the child, his parents and can also create difficult care conditions for the caregiver. These children receive multiple treatments, which is why a non-drug intervention is recommended for the management of pain and anxiety. Standard distraction (e.g.: speech) is recommended but it is often insufficient. This is why the use of interactive or hypnotic virtual reality (VR) could improve the care of these children and in particular reduce anxiety and fear. The immersion of the child in a three-dimensional environment with sound and visual stimulation potentiates the diversion of his attention. Thus, it seems necessary to evaluate the impact of interactive or hypnotic virtual reality on pain and anxiety during repeated painful care in children with acute leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Children from 6 to 16 years old suffering from leukemia requiring needle insertion into an implantable port and having a life expectancy greater than or equal to 3 months
* Subjects and their parents who have been informed of the study and having expressed their informed consent
* Children without contraindications to the use of MEOPA® :
* Patient requiring 100% oxygen ventilation
* Intracranial hypertension
* Any alteration in the state of consciousness preventing the patient's cooperation
* Children without contraindication to the use of the virtual reality mask:
* Epilepsy
* Psychiatric illness
* Children and parents able to use the self-assessment scales proposed in the study
* Enrolment in the Social Security system

Exclusion Criteria:

Children from 6 to 16:

* Having a modification of pain's integration (spina bifida for example)
* Requiring contact isolation (conjunctivitis, contagious skin condition, etc.)
* With a history of seizures

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Children's pain self-evaluation | 15 minutes after the care
  Self-evaluation of children's pain with the visual analog scale in vertical position.
  Quote from 0 to 10 with 10 being the worst score.

SECONDARY OUTCOMES:
Children's fear evaluation | 15 minutes before the care and right after the procedure
  Children's fear evaluation by the nurse with the visual analog scale from 0 to 10 with 10 being the worst score
Children's heart rate measurement | 15 minutes before the care and right after the procedure
  Heart rate mesure using a digital sensor
Evaluation of the care | After each care from the date of randomization and assessed during 3 months
  Satisfaction of the care given to the child filled out by nurses, parents and child using a questionnaire. Score going fro 1 to 3 with 3 being the best score = very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra USCLADE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (4):
- France (4):
  - CHU de Bordeaux, Bordeaux
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Assistance Publique - Hôpitaux de Marseille, Marseille
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No